CLINICAL TRIAL: NCT00108303
Title: Genetic Research in Schizophrenia Using DNA Markers and Clinical Phenotypes in Individuals Extensively Diagnosed and Genotyped
Brief Title: Genetic Research in Schizophrenia Using DNA Markers and Clinical Phenotypes
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ADRD-007-03S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dna
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic: A diagnostic was performed
  Interventions: Other: Diagnostic

INTERVENTIONS:
Other: Diagnostic — Diagnostic evaluation for schizophrenia. Schizophrenia includes schizophrenia and schizoaffective disorder.

SUMMARY:
Schizophrenia has long been known to be an illness with significant evidence for a genetic predisposition. The purpose of this study is to determine the genetic abnormalities that cause childhood and adult onset schizophrenia.

DETAILED DESCRIPTION:
It is known from genetic linkage and gene expression studies that the alpha 7 nicotinic receptor gene is abnormally expressed in people with schizophrenia. The immediate objectives of this proposal support the long-term objectives of a comprehensive description of the pathophysiology of schizophrenia and new drug treatments by carefully defining the physiological genotype-phenotype relationship for a single candidate gene. Subjects and family members with a mental illness or who appear to have a mental illness will be asked to undergo an interview, perform some mental tests and have a blood, urine, and saliva sample taken one time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals thought to have schizophrenia or schizoaffective disorder, be the parent of such an individual, or be in the matched control group of unrelated individuals not thought to have schizophrenia or schizoaffective disorder

Exclusion Criteria:

* Unable to give informed consent;
* Psychotic disorder judged to be secondary to substance abuse, psychotic disorder that appears to be secondary to a known medical or neurological disorder, or severe mental retardation

Ages: 1 Year to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Persons with schizophrenia, their relatives, and controls
Sampling Method: Non-Probability Sample
Enrollment: 538 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Freedman, MD, Principal Investigator — VA Eastern Colorado Health Care System, Denver
Locations (1):
- VA Eastern Colorado Health Care System, Denver, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Schizophrenia Probands: Persons who meet DSM-IV diagnostic criteria for schizophrenia or schizoaffective disorder.
- Schizophrenia Relatives: Subjects who are first degree relatives of subjects in Arm 1.
- Controls: Subjects who are unrelated to persons with schizophrenia and do not fulfill criteria for schizophrenia themselves.
Period: Overall Study
Arm/Group | Schizophrenia Probands | Schizophrenia Relatives | Controls
Started | 179 | 179 | 180
Completed | 179 | 179 | 180
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Schizophrenia Probands: Persons who meet DSM-IV criteria for schizophrenia or schizoaffective disorder
- Schizophrenia Relatives: Persons who are first degree relatives of persons in Arm 1
- Controls: Persons who are not related to persons in Arm 2 and do not have schizophrenia themselves.
- Total: Total of all reporting groups
Arm/Group | Schizophrenia Probands | Schizophrenia Relatives | Controls | Total
Number analyzed (Participants) | 179 | 179 | 180 | 538
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 179 | 179 | 180 | 538
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] — Age at study was taken by asking the subjects how old they were.
  years | 42 [21 to 63] | 41 [20 to 62] | 42 [20 to 63] | 42 [21 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 85 | 93 | 275
  Male | 82 | 94 | 87 | 263
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 23 | 28 | 72
  Not Hispanic or Latino | 158 | 156 | 152 | 466
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 5 | 15
  Asian | 6 | 6 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 4 | 4 | 4 | 12
  Black or African American | 40 | 41 | 40 | 121
  White | 61 | 60 | 60 | 181
  More than one race | 33 | 33 | 34 | 100
  Unknown or Not Reported | 30 | 30 | 31 | 91
Region of Enrollment [Number; unit: participants]
  United States | 179 | 179 | 180 | 538
Sensory gating ratio [Mean (Standard Deviation); unit: percent] — Ratio of the positive 50 millisecond component amplitude of the vertex auditory evoked potential in response to the second of \paired auditory tones
  percent | 68 (12) | 49 (16) | 34 (9) | 58 (12)

OUTCOME MEASURES:

1. Primary Outcome: Genetic Linkage
Description: Log of the Odds for Linkage, a standard genetic analysis metric. The number shown as a result is from a polymorphism in the promoter of the gene for the alpha7 nicotinic receptor on chromosome. Its presence in the individuals in this study, considering all three groups in one analysis, is compared to what of P50 sensory gating. P50 is a Positive wave in scalp-recorded auditory evoked potential that occurs 50 msec after the sound stimulus. P50 sensory gating is the decrement in this wave to the second of repeated sounds. The log of the odds is the common logarithm of the ratio of the odds that the gene polymorphism and P50 sensory gating are associated versus the odds that they are both distributed in the individuals at random. It is similar to the more common chi squared.
Time Frame: ten years
Population: People with schizophrenia and their relatives in families and controls as members of single families were used to establish the log of the odds ratio.
Measure: Number; unit: log (odds ratio)
Groups:
- Group 1: Subjects who receive genetic study.
Arm/Group | Group 1
Number analyzed (Participants) | 538
log (odds ratio) | 5.2
Statistical Analysis 1: Comparison: Group 1; Test type: Superiority or Other; Log (odd ratio) = 5.2
Statistical Analysis 2: Comparison: Group 1; Test type: Superiority or Other; p < 0.001, Simulation — This parameter was estimated by simulating 1000 samples with random genotypes and finding no value equal to or greater than 5.2

2. Primary Outcome: Heritability Coefficient
Description: h squared which ranges from 0 to 1. This number is similar to the more standard Pearson's correlation coefficient, except that the variable, in this case P50 sensory gating, is correlated across the statuses: schizophrenia proband (has the illness), schizophrenia relative (not ill but relative of someone who is), or control (not ill and has no known ill relative, P50 is a Positive wave in scalp-recorded auditory evoked potential that occurs 50 msec after the sound stimulus. P50 sensory gating is the decrement in this wave to the second of repeated sounds.
Time Frame: 5 years
Population: Schizophrenia probands and relatives and controls.
Measure: Number; unit: coefficient
Units Other Than Participants: Heritability
Groups:
- Schizophrenia Probands: Persons who have schizophrenia as determined by diagnosis
- Schizophrenia Relatives: Persons who are siblings or children of someone with schizophrenia
- Controls: Persons who do not have schizophrenia themselves and whose relatives do not have schizophrenia
Arm/Group | Schizophrenia Probands | Schizophrenia Relatives | Controls
Number analyzed (Participants) | 179 | 179 | 180
Number analyzed (Heritability) | 1 | 1 | 1
coefficient | 0.5 | 0.5 | 0.1
Statistical Analysis 1: Comparison: Schizophrenia Probands vs Schizophrenia Relatives vs Controls; The coefficient of segregation versus no segregation of the P50 sensory gating percent in families with schizophrenia; Test type: Superiority or Other; p = 0.001, Firsher's transform r to Z

3. Primary Outcome: Log of the ODDS of Linkage
Description: Log of the ODDS ratio of Linkage divided by the ODDS of no linkage from a maximum likelihood analysis conducted using the statistical program LINKAGE
Time Frame: 1 day
Population: Probands with schizophrenia, their relatives, and controls. The log of the odds ratio summarizes data from the entire study population.
Measure: Number; unit: units on a log scale
Groups:
- Schizophrenia Probands: Persons who meet DSM-IV diagnostic criteria for schizophrenia.
- Schizophrenia Relatives: Persons who are relatives of probands in Group 1.
- Controls: Persons who are not relatives of persons with schizophrenia and do not have schizophrenia themselves.
Arm/Group | Schizophrenia Probands | Schizophrenia Relatives | Controls
Number analyzed (Participants) | 179 | 180 | 180
units on a log scale | 5.2 | 5.2 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: People were checked for bruising at the time of study.
Groups:
- Schizophrenia Probands: Schizophrenia probands as diagnosed as having schizophrenia
- Schizophrenia Relatives: Schizophrenia relatives who siblings or children of persons with schizophrenia
- Controls: Controls who do not have personal or family history of schizophrenia
Arm/Group | Schizophrenia Probands | Schizophrenia Relatives | Controls
Serious Adverse Events (participants affected / at risk) | 0/179 | 0/179 | 0/179
Other Adverse Events (participants affected / at risk) | 0/179 | 0/179 | 0/179

LIMITATIONS AND CAVEATS:
Genetic linkage and association do not replicate well across studies. This study should be viewed in this context.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes